CLINICAL TRIAL: NCT05169983
Title: Accuracy and Feasibility of Visual Field Screening Apps - the visualFields Easy App
Brief Title: Feasibility of Visual Field Screening Apps
Acronym: VISA
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: RHM OPH0297
Record Dates: First submitted 2021-09-20; First posted 2021-12-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Visual Field Defect, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: iPad-Based Visual Field Test — In this study, the investigators aim to teach the participants to use the the visualFields easy App . The investigators will be using the app in the clinic with the patients watching, demonstrating its use and discussing and explaining its functions. Having observed how to use the application, the participant will then complete the visual field assessment.

SUMMARY:
A visual field (VF) is a measurement of how wide an area our eyes can see when fixed onto a point. Visual field testing is one of the ways of assessing how much vision there is in each eye and how much vision might have been lost over time. Defects in the visual field are seen in diseases such as glaucoma, which is one of the leading causes of blindness. VF tests should be performed regularly during outpatient appointments to help monitor these conditions before they progress. Monitoring individuals with VF defects presents a large strain on eye services at University Hospitals Southampton (UHS).

Recently an Apple iPad-based application called 'VisualFields easy' has been developed that could be used at home to test visual fields, opening up the possibility of remote monitoring. This is especially significant since the onset of the COVID-19 pandemic which has left outpatient clinics across the UK with large patient backlogs. However, it's not understood yet to what level of accuracy this iPad test can be performed by untrained people and whether the results of this test are medically reliable.

This study will measure if there's a correlation between iPad-based VF measurements and the standard clinic-based measurements taken by professionals. The potential of this app to be used at home will also be assessed with a usability questionnaire. These measurements will be taken during routine eye and neurology outpatient clinics at UHS. Home-based VF testing could allow those who weren't able to access eye services during the pandemic greater follow-up and monitoring. Through providing regular, up-to-date information on a patient's condition and progress, VF tests at home may improve outcomes. The investigators also foresee the benefits of this app on NHS clinical services, with the potential of reduced outpatient appointments and waiting times thus easing pressure on the NHS.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 17 or older
* Familiar with and able to use tablet technology

Exclusion Criteria:

* Patient not willing to participate in the study and give written informed consent
* Patients with learning difficulties that preclude reliable assessment of visual fields

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants will be recruited from the ophthalmology and neurology outpatient clinics in Southampton General Hospital. Typically, patients in these clinics are seen for a variety of ocular and neurological diagnoses and will be undergoing visual field testing as part of their routine care.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Accuracy of the visualFields easy App | Through study completion, an average of 1 year
  To determine the statistical strength and / or presence or absence of correlation between the iPad-based visual field assessment procedure in comparison to clinic-based visual field assessment.

SECONDARY OUTCOMES:
Feasibility of home-based visual field assessment | Through study completion, an average of 1 year
  To explore through a quantitative questionnaire, the possible feasibility and utility of home-based visual field assessment

CONTACTS AND LOCATIONS:
Overall Officials: Helena Lee, PhD, Principal Investigator — Associate Professor & Honorary Consultant Ophthalmologist
Locations (1):
- Eye Unit, University Hospitals Southampton NHS Foundation Trust, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No